CLINICAL TRIAL: NCT04273269
Title: An Open-Label Adaptive-Design Study of Intracisternal Adenoassociated Viral Vector Serotype rh.10 Carrying the Human β-Galactosidase cDNA for Treatment of GM1 Gangliosidosis
Brief Title: A Safety and Efficacy Study of LYS-GM101 Gene Therapy in Patients With GM1 Gangliosidosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The clinical trial is closed due to Lysogene's cessation of activities. This study closure is not due to safety reasons.
Sponsor: LYSOGENE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1-GM-101
Record Dates: First submitted 2020-01-21; First posted 2020-02-18 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: GM1 Gangliosidosis
Keywords: GM1 Gangliosidosis; Lysosomal Storage Disease; Landing Disease
MeSH Terms: conditions — Gangliosidosis, GM1; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 8x10^12 vg/Kg LYS-GM101 (Experimental): Subjects will receive a single infusion: 8x10^12 vg/Kg LYS-GM101
  Interventions: Genetic: LYS-GM101

INTERVENTIONS:
Genetic: LYS-GM101 — LYS-GM101 is an adeno-associated viral vector serotype rh.10 (AAVrh.10) carrying the human β-galactosidase gene, formulated as a suspension for injection

SUMMARY:
LYS-GM101 is a gene therapy for GM1 gangliosidosis intended to deliver a functional copy of the GLB1 gene to the central nervous system. This study will assess, in a 2-stage adaptive-design, the safety and efficacy of treatment in subjects with infantile GM1 gangliosidosis.

DETAILED DESCRIPTION:
GM1 gangliosidosis is a fatal autosomal recessive disease caused by mutations in the GLB1 gene leading to accumulation of GM1 ganglioside in neurons and progressive neurodegeneration. There are three pediatric subtypes: early infantile, late infantile and juvenile. This is an interventional, multicenter, single-arm, 2-stage adaptive design study of LYS-GM101 for which the first stage (Stage 1) is for safety evaluation (FIH) and the second stage (Stage 2) will establish efficacy as compared to the natural history of the disease. The participants with infantile GM1 gangliosidosis will receive a single dose of LYS-GM101 by intracisternal injection. After a two-year evaluation period (main part of the study), each participant will be followed for an additional three-year long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Documented GM1 gangliosidosis diagnosis based on genotyping confirming the β-gal gene mutations and/or documented deficiency of β-gal enzyme by laboratory testing
* Children with early infantile GM1 gangliosidosis less than 12 months of age with ability to swallow
* Children with late infantile GM1 gangliosidosis less than 3 years of age with ability to sit

Exclusion Criteria:

* Uncontrolled seizure disorder. Patients who are stable on anti-convulsive medications may be included
* More than 40% brain atrophy as measured by MRI total brain volume at screening
* Current participation in a clinical trial of another investigational medicinal product
* Past participation in a gene therapy trial
* History of hematopoietic stem cell transplantation
* Any condition that would contraindicate treatment with immunosuppressant therapy
* Presence of concomitant medical condition or anatomical abnormality precluding lumbar puncture or intracisternal injection
* Presence of any permanent items (e.g., metal braces) precluding undergoing MRI
* History of non-GM1 gangliosidosis medical condition that would confound scientific rigor or interpretation of results
* Rare and unrelated serious comorbidities, e.g., Down syndrome, intraventricular hemorrhage in the new-born period, extreme low birth weight (<1500 grams) or known bleeding disorders
* Any vaccination 1 month prior to the planned immunosuppressant treatment
* Serology consistent with HIV exposure or consistent with active hepatitis B or C infection
* Grade 2 or higher lab abnormalities for Liver function tests (LFT), bilirubin, creatinine, hemoglobin, white blood cell (WBC) count, platelet count, prothrombin time (PT), and partial thromboplastin time (PTT), according to CTCAE v5.0

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Stage 1: Physical examination by body system | Up to 6 months (multiple visits)
  Physical examination by body system: normal/abnormal and change from previous assessment
Stage 1: Neurological examination | Up to 6 months (multiple visits)
  Neurological examination: normal/abnormal motor activity and coordination, and change from previous assessment
Stage 1: Vital signs: change from baseline in heart rate | Up to 6 months (multiple visits)
  Vital signs: change from baseline in heart rate
Stage 1: Vital signs: change from baseline in body temperature | Up to 6 months (multiple visits)
  Vital signs: change from baseline in body temperature
Stage 1: Vital signs: change from baseline in diastolic and systolic blood pressure | Up to 6 months (multiple visits)
  Vital signs: change from baseline in diastolic and systolic blood pressure
Stage 1: Imaging: presence of bleeding post-administration | Up to 6 months (multiple visits)
  Imaging: presence of bleeding post-administration
Stage 1: Change from baseline in biochemistry laboratory parameters | Up to 6 months (multiple visits)
  Change from baseline in biochemistry laboratory parameters
Stage 1: Change from baseline in coagulation and hematology laboratory parameters | Up to 6 months (multiple visits)
  Change from baseline in coagulation and hematology laboratory parameters
Stage 1: Incidence of treatment-emergent adverse event and serious adverse events | Up to 6 months (multiple visits)
  Incidence of treatment-emergent adverse event and serious adverse events
Stage 1: Assessment of humoral immune response by measurement of antibodies anti-AAV and anti-beta-galactosidase (ELISA) and cellular immune response by beta-galactosidase-specific T-cell proliferation assay | Up to 6 months (multiple visits)
  Assessment of humoral immune response by measurement of antibodies anti-AAV and anti-beta-galactosidase (ELISA) and cellular immune response by beta-galactosidase-specific T-cell proliferation assay

SECONDARY OUTCOMES:
Motor Function | Up to 2 years (multiple visits)
  Assess change from baseline in motor function using the Hammersmith Infant Neurological Evaluation (HINE) or Hammersmith Functional Motor Scale-Expanded (HFMSE) instruments
Brain MRI | Up to 2 years (multiple visits)
  Assess brain atrophy and brain volume
Developmental changes (VABS-II) | Up to 2 years (multiple visits)
  Assess developmental change from baseline in the Vineland Adaptive Behavior Scale-II-Expanded Interview (VABS-II) instrument
Developmental changes (BSID-III or KABC-II) | Up to 2 years (multiple visits)
  Assess developmental change from baseline in the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or the Kaufman Assessment Battery for Children, 2nd Edition (KABC-II) instruments
Blood and cerebrospinal fluid (CSF) biomarkers (beta-galactosidase) | Up to 2 years (multiple visits)
  Assess change in beta-galactosidase activity measured from baseline
Blood and cerebrospinal fluid (CSF) biomarkers (GM1 ganglioside) | Up to 2 years (multiple visits)
  Assess change in GM1 ganglioside level measured from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — LYSOGENE
Locations (3):
- Children's Hospital of Orange County (CHOC), Orange, California, United States
- Hôpital Armand-Trousseau, Centre de Référence des Maladies Lysosomales (CRML), Service de Neuropédiatrie, Paris, France
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739